CLINICAL TRIAL: NCT02352480
Title: A Multi-Center, Prospective, Randomized Trial Comparing the Effectiveness of Aurix Therapy to Usual and Customary Care in All Wagner Grades of Diabetic Foot Ulcers
Brief Title: Effectiveness of Aurix Therapy in Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nuo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM002 Gold
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Diabetic Foot Ulcers
Keywords: Non Healing Wound
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aurix + UCC (Experimental): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive Aurix treatment plus usual and customary care, which can include any advanced therapeutics.
  Interventions: Device: Aurix
- Usual and Customary Care (No Intervention): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week there after while receiving usual and customary care, but actual frequency of visits will be determined by the treating physician. Usual and customary care, which can include any advanced therapeutics.

INTERVENTIONS:
Device: Aurix — Aurix is a platelet-rich plasma (PRP) gel used in the treatment of non-healing chronic wounds. It will be administered twice weekly for 2 weeks then weekly.
  Arms: Aurix + UCC

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, randomized trial in which diabetic food ulcers (DFU) will be treated using Aurix plus Usual and Customary Care (UCC) and compared to a group receiving just UCC as provided in up to 100 U.S. wound centers

DETAILED DESCRIPTION:
Aurix is a platelet-rich plasma gel used in the treatment of non-healing chronic wounds. Prospective observational studies of the effectiveness of Aurix have demonstrated promising results in regard to the healing of DFUs, including severe Wagner grade 3 and 4 ulcers. The aim of this trial is to demonstrate the of complete wound healing in a prospective, open-label, randomized trial in which diabetic foot ulcers will be treated using Aurix to determine the time to heal at 12 weeks. Comparison will be made on a 1:1 basis of Aurix + UCC versus control subjects receiving undefined UCC.

ELIGIBILITY:
Inclusion Criteria:

1. Medicare eligible
2. ≥18 years of age
3. Type I or II diabetes requiring medical treatment as determined by the physician
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) is a Wagner 1-5 DFU (see Appendix 9 for Wagner Classification) that is located on the dorsal, plantar, medial, or lateral aspect of the foot or heel (including all toe surfaces)
5. For subjects with potentially multiple eligible DFUs, the largest ulcer will be selected as the Index Ulcer for study. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 0.5 cm2 and 50 cm2
7. Subject has received UCC care for ≥ 2 weeks at treating wound clinic
8. Demonstrated adequate offloading regimen
9. Duration ≥ 1 month at first visit
10. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to Aurix components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Presence of another wound that is concurrently treated and might interfere with treatment of the index wound by Aurix
3. Ulcer not of DFU pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
4. Patients on chemotherapeutic agents or any malignancy in the wound area
5. Subjects who are cognitively impaired
6. Serum albumin of less than 2.5 g/dL
7. Plasma Platelet count of less than 100 x 109/L
8. Hemoglobin of less than 10.5 g/dL
9. Subject has inadequate venous access for repeated blood draw required for Aurix administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Time to heal | 12 weeks
  The primary endpoint of the trial is determine the time to heal diabetic foot ulcers treated with Aurix and Standard of Care at 12 weeks. Comparison will be made with the control arm of subjects treated only with Standard of Care.

SECONDARY OUTCOMES:
Incidence of amputations | 12 weeks
  Frequency of lower extremity amputations; major/minor amputations will be tabulated but not tested.
Proportion of completely healed ulcers | 12 weeks
  Proportion of patients with completely healed diabetic foot ulcers
W-QOL (Quality of life with chronic wounds) score | 12 weeks
  Change in mean W-QOL (Quality of life with Chronic Wounds) score between baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clausen, PhD, Study Director — Nuo Therapeutics
Locations (20):
- United States (20):
  - Methodist Hospital Wound Care Center, Arcadia, California
  - Beverly Hospital Wound and Hyperbaric Center, Montebello, California
  - Kaweah Delta Rehabiliation Hospital, Visalia, California
  - Bristol Hospital Wound Care Center, Bristol, Connecticut
  - Piedmont, Atlanta, Georgia
  - St. Luke's Wound and Hyperbaric Center, Meridian, Idaho
  - The Center for Wound Healing at FHN, Freeport, Illinois
  - Tufts Medical Center - Center for Wound Healing, Boston, Massachusetts
  - St Joseph Mercy Oakland Hospital Center for Wound Care and Hyperbaric Medicine, Pontiac, Michigan
  - Catskill Regional Medical Center - Wound Healing Center, Harris, New York
  - Orange Regional, Middletown, New York
  - The Wound Center of Niagara, Niagara Falls, New York
  - Onslow Memorial Hospital - Wound Care and Hyperbaric Center, Jacksonville, North Carolina
  - The Center for Wound Healing Crozer Chester Medical Center, Chester, Pennsylvania
  - Memorial Hermann Memorial City, Houston, Texas
  - Memorial Hermann South West, Houston, Texas
  - Memorial Hermann South East, Houston, Texas
  - Memorial Hermann Katy Rehab, Katy, Texas
  - St. Mary's Wound and Hyperbaric Center, Huntington, West Virginia
  - The Center for Wound Healing Cabell Huntington Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No